CLINICAL TRIAL: NCT04100057
Title: Sleep Disturbance and Emotion Regulation Brain Dysfunction as Mechanisms of Neuropsychiatric Symptoms in Alzheimer's Dementia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Andrea Goldstein-Piekarski, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-53039; R01MH120776 (NIH)
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Neuropsychiatric Symptoms; Sleep Disturbance
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Parasomnias | interventions — Cognitive Behavioral Therapy; Desensitization, Psychologic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy for Insomina (CBT-I) (Experimental): CBT-I improves sleep through a combination of behavioral interventions (stimulus control (SC), sleep restriction (SR)), cognitive therapy (CT) as well as additional components such as mindfulness training and sleep hygiene education. SC is an intervention that re-establishes the connection between the bed/bedroom with sleep to help develop a more consistent sleep/wake pattern. SR leads to higher quality sleep by reducing excessive time spent in bed to the actual amount of sleep, thereby creating mild sleep deprivation and increasing the homeostatic sleep drive. Like CT for other disorders, CT for insomnia targets maladaptive thoughts and cognitions that may interfere with sleep.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I)
- Desensitization Therapy for Insomnia (DT-I) (Active Comparator): DT-I is a quasidesensitization treatment presented as a means of eliminating the "conditioned arousal," which prolongs nocturnal awakenings. DT-I has been validated as an active-placebo control condition. Therapists help each DT-I recipient develop a chronological 12-item hierarchy of common activities he/she does on awakening at night (e.g., opening eyes, clock watching). Therapists also help them develop 6 imaginal scenes of themselves engaged in neutral activities (e.g., reading the newspaper). Each session, DT-I recipients are taught to pair neutral scenes with items on the 12-item hierarchy so, by the end of the sixth session, all hierarchy items have been practiced with therapist assistance. Each session, the exercise is tape recorded and the patient is given this tape locked in a player. The patients are told to practice their exercises at home once each day, no less than 2 hours before bedtime, but to avoid using the tape or exercise during sleep periods.
  Interventions: Behavioral: Desensitization Therapy for insomnia (DT-I)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I) — CBT-I improves sleep through a combination of behavioral interventions (stimulus control (SC), sleep restriction (SR)), cognitive therapy (CT) as well as additional components such as mindfulness training and sleep hygiene education. SC is an intervention that re-establishes the connection between the bed/bedroom with sleep to help develop a more consistent sleep/wake pattern. SR leads to higher quality sleep by reducing excessive time spent in bed to the actual amount of sleep, thereby creating mild sleep deprivation and increasing the homeostatic sleep drive. Like CT for other disorders, CT for insomnia targets maladaptive thoughts and cognitions that may interfere with sleep.
  Arms: Cognitive Behavioral Therapy for Insomina (CBT-I)
Behavioral: Desensitization Therapy for insomnia (DT-I) — DT-I is a quasidesensitization treatment presented as a means of eliminating the "conditioned arousal," which prolongs nocturnal awakenings. DT-I has been validated as an active-placebo control condition. Therapists help each DT-I recipient develop a chronological 12-item hierarchy of common activities he/she does on awakening at night (e.g., opening eyes, clock watching). Therapists also help them develop 6 imaginal scenes of themselves engaged in neutral activities (e.g., reading the newspaper). Each session, DT-I recipients are taught to pair neutral scenes with items on the 12-item hierarchy so, by the end of the sixth session, all hierarchy items have been practiced with therapist assistance. Each session, the exercise is tape recorded and the patient is given this tape locked in a player. The patients are told to practice their exercises at home once each day, no less than 2 hours before bedtime, but to avoid using the tape or exercise during sleep periods.
  Arms: Desensitization Therapy for Insomnia (DT-I)

SUMMARY:
Recent findings suggest that sleep disruption may contribute to the generation and maintenance of neuropsychiatric symptoms including anxiety, depression, agitation, irritation, and apathy while treating sleep disruption reduces these symptoms. Impairments in the neural systems that support emotion regulation may represent one causal mechanism mediating the relationship between sleep and emotional distress. However, this model has not yet been formally tested within a sample of individuals with or at risk for developing Alzheimer's Disease (AD)

This proposal aims to test a mechanistic model in which sleep disturbance contributes to neuropsychiatric symptoms through impairments in fronto-limbic emotion regulation function in a sample of individuals at risk for developing, or at an early stage of AD.

This study seeks to delineate the causal association between sleep disruption, fronto-limbic emotion regulation brain function, and neuropsychiatric symptoms. These aims will be achieved through a mechanistic, randomized 2-arm controlled trial design. 150 adults experiencing sleep disturbances and who also have cognitive impairment with the presence of at least mild neuropsychiatric symptoms will be randomized to receive either a sleep manipulation (Cognitive Behavioral Therapy for Insomnia CBT-I; n=75) or an active control (n=75). CBT-I improves sleep patterns through a combination of sleep restriction, stimulus control, mindfulness training, cognitive therapy targeting dysfunctional beliefs about sleep, and sleep hygiene education. Neuropsychiatric symptoms, fronto-limbic functioning, and sleep disruption will be assessed at baseline and at the end of the sleep manipulation through functional Magnetic Resonance Imaging (fMRI), clinical interviews, PSG recordings, and self-report questionnaires. Neuropsychiatric symptoms (anxiety and depression) and sleep disturbance (actigraphy, Insomnia Severity Index, and sleep diaries) will be assayed at baseline and each week throughout the sleep manipulation to assess week-to-week changes following an increasing number of CBT-I sessions. Wristwatch actigraphy will be acquired from baseline to the end of the sleep manipulation at week 11. Neuropsychiatric symptoms and sleep will be assessed again at six months post-manipulation.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of any racial or ethnic group, aged 50-90 (inclusive)
* Subjective complaint of insomnia associated with daytime impairment or distress (ISI ≥ 10)
* Subjective complaint of sleep disturbance ≥ 3 months in duration
* Subjective complaint of Neuropsychiatric symptoms (Self-Report NPI distress total score ≥ 4 on any measure other than the sleep domain OR current symptoms from Study Partner NPI ≥ 1
* Able to verbalize understanding of involvement in the research and provide written informed consent or provide assent co-signed by a LAR
* Fluent and literate in English
* Written, informed consent
* Medications (including any dementia-related meds) stable for at least 4 weeks prior to study baseline
* Research diagnosis of memory impairment based on the following:

  i) Global Clinical Dementia Rating (CDR) of 0.5 or 1.0. OR a diagnosis of memory impairment from the Stanford/VA AD Center
* MRI safety screen passed , as assessed by the attached MRI safety screening form from the Stanford CNI, excluding mild claustrophobia that will be further screened at the in-person screening session per the screening protocol
* Have a caregiver or study partner willing to aid in facilitating the protocol and ratings
* Reside within approximately 60 miles of Stanford University

Exclusion Criteria:

* less than 20 on the Mini-Mental State Examination (MMSE)
* Acute or unstable chronic illness: including but not limited to: uncontrolled thyroid disease, kidney, prostate or bladder conditions causing excessively frequent urination (> 3 times per night); medically unstable congestive heart failure, angina, other severe cardiac illness as defined by treatment regimen changes in the prior 3 months; stroke with serious sequelae; cancer if < 1 year since end of treatment; asthma, emphysema, or other severe respiratory diseases uncontrolled with medications; and neurological disorders (with the exception of mild AD) such as Parkinson's disease and unstable epilepsy as defined by treatment regimen changes in the prior 3 months; unstable adult onset diabetes as defined by treatment regimen changes in the prior 3 months.
* Use of medication specifically prescribed for sleep disturbance or nighttime-only, low dose anti-depressants (e.g., doxepin, amitriptyline, trazodone used only at sub-therapeutic anti-depressant doses and taken only at bedtime) specifically prescribed for sleep disturbance and unwilling or unable to discontinue > two weeks (anti-depressants) or >1 week (sleep medications) prior to baseline data collection.
* Current or lifetime history of bipolar disorder
* History of psychosis preceding onset of memory impairments
* Substance abuse or dependence
* Excessive alcohol consumption (>14 drinks per week or > 4 drinks per occasion)
* Current exposure to trauma, or exposure to trauma within the past 3 months
* Presence of suicidal ideations representing high risk as measured by the Columbia-Suicide Severity Rating Scale (C-SSRS). Individuals are considered high risk if they have endorsement of either of the following:

  1. A score of 4 or more for the past month on the C-SSRS
  2. ) A positive endorsement, relative to the past 90 days, in the "Suicide Behavior" section of item #6 (Have you ever done anything, started to do anything, or prepared to do anything to end your life?)
* History of significant head trauma followed by persistent neurologic deficits or known structural brain abnormalities OR traumatic brain injury in the past two months
* Severe impediment to vision, hearing and/or hand movement, likely to interfere with the ability to complete the assessments, or are unable and/or unlikely to follow the study protocols
* Current or expected cognitive behavior therapy or other evidence based psychotherapies; therapy for another condition (e.g. Depression)
* History of falling and/or severe mobility impairment
* Individuals who are not CPAP adherent or have untreated severe OSA (AHI >= 30).CPAP adherence being defined as using the CPAP machine 70% of nights for a minimum of 4 hours per night.
* Received Cognitive Behavior Therapy for Insomnia (CBT-I) or Desensitization Therapy for Insomnia (DTI) within the past year
* Are not fully vaccinated for COVID-19 (e.g. 2 doses of Moderna or BioNTech, Pfizer vaccines; or 1 for Johnson and Johnson) and unwilling, if asked, to provide proof (e.g., CDC COVID-19 Vaccination Card, e-Health record, etc.)

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Fronto-limbic function | change between baseline and 6 weeks
  Fronto-limbic function will be assessed through functional magnetic resonance imaging.
Neuropsychiatric Symptoms | 6 weeks
  The Neuropsychiatric Inventory Questionnaire (NPI) examines 12 sub-domains of behavioral functioning. We will be using a summed composite score of 7 domains (agitation/aggression, dysphoria, anxiety, euphoria, apathy, disinhibition, and irritability/lability) as the primary outcome measure as these domains have been most closely related to sleep disturbance. Severity of symptoms for each domain are rated on a scale of 0 - 3 (Higher scores indicate greater Severity). The overall summed composite score will be created by summing the total score for each of the 7 domains of interest. This will yield an overall summed composite score ranging from 0 to 21 (higher scores indicate worse symptoms). This questionnaire will be administered as self report to the participant as well as an informant to the study partner.
Insomnia symptoms | 6 weeks
  The participant's subjective experience of severity of insomnia using the Insomnia Severity Index (ISI). The ISI has been shown to be a reliable subjective measure of insomnia severity as well as a sensitive measure of symptom change. Recently it has also been related to objective polysomnography measures. The scale ranges from 0 to 28, with a score of 0-7 indicating no clinically significant insomnia, scores 8-14 indicating sub threshold insomnia, 15-21 indicating moderate insomnia and 22-28 indicating severe insomnia.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Goldstein-Piekarski, PhD, Principal Investigator — Stanford University
Locations (1):
- Andrea Goldstein-Piekarski, PhD, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No